CLINICAL TRIAL: NCT04822337
Title: A Phase I/II Study of Carfilzomib, Lenalidomide, Dexamethasone and the Anti-B-Cell Maturation Antigen (BCMA) Antibody Drug Conjugate Belantamab Mafodotin in Multiple Myeloma
Brief Title: Study of Carfilzomib, Lenalidomide, Dexamethasone and Belantamab Mafodotin in Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Amgen (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00081609; Pro00050160 (Other: Advarra IRB); LCI-HEM-NDMYE-KRDB-001 (Other: Atrium)
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Plasma Cell Neoplasms; BCMA
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — carfilzomib; Lenalidomide; Dexamethasone; belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): Carfilzomib, Lenalidomide, Dexamethasone, Belantamab Mafodotin
  Interventions: Drug: Carfilzomib, Lenalidomide, Dexamethasone, Belantamab Mafodotin
- Phase II (Experimental): Carfilzomib, Lenalidomide, Dexamethasone, Belantamab Mafodotin
  Interventions: Drug: Carfilzomib, Lenalidomide, Dexamethasone, Belantamab Mafodotin

INTERVENTIONS:
Drug: Carfilzomib, Lenalidomide, Dexamethasone, Belantamab Mafodotin — Phase I - Chemotherapy multiple agents systemic Phase II - Maximum Tolerated Dose from Phase I

SUMMARY:
This research study is being done to learn if the study drug belantamab mafodotin, in combination with other standard medications, can improve multiple myeloma. This study will also help determine what effects, good and/or bad, this combination of study drugs have on subjects and their cancer, and to evaluate the overall response to this study treatment combination.

DETAILED DESCRIPTION:
This is a phase I dose escalation and expansion study in RMM and RRMM followed by a single arm phase II expansion in high risk, NDMM. The phase I portion of the protocol will utilize a standard 3+3 dose escalation design to determine the maximum tolerated dose (MTD) and RP2D of the KRd-belantamab mafodotin combination. The phase II portion of the trial is a two-stage design that will assess the efficacy and safety of the combination in newly diagnosed, high-risk MM patients.

ELIGIBILITY:
INCLUSION CRITERIA for all subjects:

1. Written informed consent and HIPAA authorization for release of personal health information signed by the subject or his/her legally authorized representative. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age greater than or equal to 18 years at the time of consent. Because no dosing or adverse event data are currently available on the use of belantamab mafodotin as a single agent or in combination with KRd in subjects less than 18 years of age, children are excluded from this study.
3. ECOG Performance Status of less than or equal to 2
4. Demonstrate adequate organ function
5. Adequate cardiac function as defined by a greater than 40% left ventricular ejection fraction (LVEF) by ECHO, cardiac MRI or MUGA

   1. Note for subjects in phase II: if a cycle of pre-study induction therapy containing a PI or anthracycline was administered, assessment of the LVEF must be repeated.
6. For those with symptomatic pulmonary disease with Grade 2 or higher symptoms (e.g. COPD, asthma) or other signs / symptoms of pulmonary disease, adequate pulmonary function as defined by a FEV1 greater than or equal to 50% of predicted and DLCO/VA greater than or equal to 50% of predicted
7. Females of childbearing potential (FCBP) must have two negative serum pregnancy tests during screening: the first within 10-14 days prior to first dose of study treatment and the second within 24 hours prior to first dose of study treatment. NOTE: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), are amenorrhoeic for less than 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation; or are postmenopausal (at least 12 consecutive months with no menses without an alternative medical cause).
8. FCBP must be willing to use 2 effective contraceptive methods (at least one that is highly effective) or abstinence starting from the time of informed consent, while on belantamab mafodotin and lenalidomide. If either drug is discontinued, 2 effective forms of contraception should be continued until at least 4 weeks after the last dose of lenalidomide, and 1 form of effective contraception should be continued until 4 months post last dose of belantamab mafodotin. FCBP should use effective contraception or abstinence from consent until 30 days after last treatment with carfilzomib, and males with a partner of childbearing potential must use effective contraception or abstinence for at least 90 days post last dose of carfilzomib.
9. Male subjects must agree to the following from the first dose of study treatment until 6 months after the last dose of belantamab mafodotin, to allow for clearance of altered sperm:

   1. Refrain from donating sperm

      PLUS either:
   2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent. OR
   3. Must agree to use effective contraception/barrier as detailed below:

      Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner of reproductive potential to use an additional highly effective contraceptive method with a failure rate of less than 1% per year
10. FCBP must agree not to donate eggs (ova, oocytes) for the purpose of reproduction during the intervention period and for at least 4 months after the last dose of study intervention belantamab mafodotin, at least 30 days after the last dose of carfilzomib, and at least 4 weeks after the last dose of lenalidomide.
11. As determined by the enrolling physician, ability of the subject to understand and adhere with study procedures for the entire length of the study
12. Ability to swallow oral medications
13. Willing to refrain from using contact lenses while participating in this study

INCLUSION CRITERIA - Phase I treatment for Relapsed or Relapsed/Refractory MM:

1. Subjects with Relapsed or Relapsed/Refractory MM who have had at least 1 line of prior therapy.

   1. Refractory is defined as less than 25% reduction in M-protein or progression of disease during treatment or within 60 days after cessation of treatment
   2. A line of therapy is defined as one or more cycles of a planned treatment program.

      This may consist of one or more planned cycles of single-agent therapy or combination therapy, as well as a sequence of treatments administered in a planned manner. A new line of therapy starts when a planned course of therapy is modified to include other treatment agents (alone or in combination) as a result of disease progression, relapse, or toxicity. A new line of therapy also starts when a planned period of observation off therapy is interrupted by a need for additional treatment for the disease.
2. Subjects must have measurable disease, as defined by at least one of the following:

   1. Serum monoclonal protein level greater than or equal to 0.5 g/dL
   2. 24-hour urinary M-protein greater than or equal to 200 mg
   3. Involved free light chain level greater than or equal to 10 mg/dL, along with an abnormal free light chain ratio (defined as less than 0.26 or greater than 1.65).
3. Subject must have not progressed on full dose lenalidomide previously (25 mg on days 1-21 of a 28-day cycle or its dosing equivalent based on renal function at the time of progression)
4. Prior to enrollment:

   a. There should be a washout period of ≥14 days from any prior chemotherapy AND b. The subject must have adequate recovery from toxicity of prior chemotherapy as defined by the following: i. Hematologic lab results within parameters noted in Table 3.2.1 ii. Non-hematologic toxicity resolved to grade 1 or baseline with the following exceptions:

<!-- -->

1. Subjects who have started a course of antibiotic therapy for infection and symptoms have improved to baseline or grade 1, but remain on antibiotic therapy are eligible
2. Subjects with ≤grade 2 fatigue are eligible
3. Subjects with ≤grade 2 hyperglycemia are eligible, even if pharmacologic treatment was required
4. Subjects with ≤grade 2 electrolyte abnormalities are eligible, even if pharmacologic treatment was required
5. Subjects with ≤grade 2 nausea, constipation or diarrhea are eligible, even if pharmacologic treatment was required
6. Subjects with less than grade 2 peripheral neuropathy

INCLUSION CRITERIA - Phase II treatment for high-risk newly diagnosed MM:

1. Active, newly diagnosed multiple myeloma with CRAB features or a myeloma-defining event per the IMWG 2014 criteria. Note: It is acceptable to include subjects who have had one cycle of emergent treatment for multiple myeloma.
2. High-risk disease, as defined by at least one of the following:

   i. Del(1p) ii. Gain of 1q21 [greater than or equal to 3 copies] iii. Monosomy 13 or del(13q) by conventional karyotype iv. High risk IgH translocation [t(4;14), t(14;16) or t(14;20)] v. del(17p)
3. Measurable disease by 1 or more of the following:

   a. Serum monoclonal protein level greater than or equal to 0.5 g/dL b. 24-hour urinary M-protein greater than or equal to 200 mg c. Involved free light chain level greater than or equal to 10 mg/dL (100 mg/L), along with an abnormal free light chain ratio (defined as less than 0.26 or greater than 1.65).

   d. Note: for subjects who have received a prior cycle of non-protocol therapy, measurable disease will be based on the serum and urine monoclonal protein and serum free light chain levels prior to the cycle of non-protocol therapy
4. No more than one prior cycle of non-protocol therapy will be allowed, recognizing that high-risk multiple myeloma subjects frequently require immediate therapy at initial diagnosis even before risk assessment is complete. For those subjects who receive a cycle of non-protocol induction therapy:

   a. There should be a washout period of ≥14 days from the last dose of pre-study therapy AND b. The subject must have adequate recovery from toxicity of pre-study therapy as defined by the following: i. Hematologic lab results within parameters ii. Non-hematologic toxicity resolved to grade 1 or baseline with the following exceptions:

1. Subjects who have started a course of antibiotic therapy for infection and symptoms have improved to baseline or grade 1, but remain on antibiotic therapy are eligible 2. Subjects with less than or equal to grade 2 fatigue are eligible 3. Subjects with less than or equal to grade 2 hyperglycemia are eligible, even if pharmacologic treatment was required 4. Subjects with less than or equal to grade 2 electrolyte abnormalities are eligible, even if pharmacologic treatment was required 5. Subjects with less than or equal to grade 2 nausea, constipation or diarrhea are eligible, even if pharmacologic treatment was required 6. Subjects with less than grade 2 peripheral neuropathy

EXCLUSION CRITERIA for all subjects:

1. Active infection requiring systemic therapy. NOTE: at the discretion of the treating investigator, subjects who have started antibiotic therapy for subjects who had symptoms present, symptoms must have improved to baseline or grade 1 in severity may start treatment prior to completion of their course of antibiotic therapy.
2. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study.)
3. Subjects cannot have other prior or concomitant malignancies except for:

   1. Curatively treated non-melanoma skin cancer
   2. Other cancer for which the subject has been medically stable for at least 2 years and/or, in the opinion of the Site Principal Investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy
4. Active central nervous system (CNS) involvement
5. Concomitant AL amyloidosis or POEMS syndrome
6. Plasma cell leukemia
7. Treatment with any investigational drug within 14 days or five half-lives, whichever is shorter, prior to first dose of study treatment.
8. Medical, psychiatric, or other condition/disorder (including lab abnormalities) which, in the opinion of the treating physician, would make this protocol treatment unreasonably hazardous for the subject, or could interfere with obtaining informed consent or compliance to the study procedures
9. Significant cardiac disease, including any of the following:

   1. Greater than or equal to Class 3 New York Heart Association (NYHA) congestive heart failure (see Appendix B)
   2. ECG evidence of acute ischemia
   3. Unstable angina
   4. Myocardial infarction, Coronary angioplasty, stenting, or bypass grafting within three months prior to day 1 of treatment
   5. Clinically significant uncontrolled and/or untreated arrhythmias or conduction block, including clinically significant ECG abnormalities such as 2nd degree Mobitz Type ll or 3rd degree atrioventricular (AV)block. However, PACs, PVCs, rate controlled atrial fibrillation, sinus arrhythmia, asymptomatic sinus bradycardia or sinus tachycardia and 1st degree heart block are not considered clinically significant.
   6. Greater than or equal to Grade 2 QTcF prolongation (i.e. >480 msec)
10. Uncontrolled hypertension, defined as a systolic blood pressure of greater than or equal to 160 mmHg or a diastolic blood pressure of greater than or equal to 90 mmHg
11. Grade greater than or equal to 2 peripheral neuropathy
12. Psychiatric illness/social situation that would limit compliance with study requirements as determined by the investigator
13. Known immediate or delayed hypersensitivity or allergic reaction to any components of, or related to, protocol therapy (e.g. during exposure to carfilzomib, lenalidomide or dexamethasone as part of a pre-study cycle of therapy).
14. History of erythema multiforme to lenalidomide or other IMID
15. Discontinuation of prior carfilzomib, lenalidomide or dexamethasone due to treatment toxicity
16. Major surgery within 4 weeks prior to day 1 of treatment
17. Radiation within 14 days prior to day 1 of treatment. Note: palliative XRT to less than 5% of the total marrow volume as assessed by the treating investigator is allowed within 14 days prior to day 1 of treatment
18. Current corneal epithelial disease except mild changes in corneal epithelium
19. Positive hepatitis C antibody test result (this test preferable) or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment

    a. NOTE: Subjects with positive Hepatitis C antibody due to prior eradicated disease can be enrolled if a confirmatory negative Hepatitis C RNA test is obtained
20. A known diagnosis of HIV
21. Is seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e. subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Subjects who are PCR positive will be excluded. Subjects with Hepatitis B surface antibodies and previous Hepatitis B vaccination will be eligible.
22. Has current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria
23. Participant must not have presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided they fulfill inclusion criteria
24. Participant must not have had plasmapheresis within 7 days prior to first dose of study treatment
25. Any evidence of active mucosal or internal bleeding
26. Participant must not be simultaneously enrolled in any therapeutic clinical trial
27. Administration of live or live-attenuated vaccines within 30 days prior to the first dose of study treatment

    a. Exception: Monkeypox vaccine may be given if there are at least 3 days between the vaccine and initiation of study treatment.
28. Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Establish Maximum Tolerated Dose (MTD) | time to complete Cycle 1 (28 days)
  DLTs will be determined for each subject enrolled in Phase I as a binary variable indicating whether the subject experienced a DLT during Cycle 1 of belantamab mafodotin-containing protocol directed induction therapy.
Evaluate Complete Response (CR) | up to 5 years
  CR will be determined for each subject as a binary variable indicating whether the achieved a best overall response to induction therapy of CR or better.

SECONDARY OUTCOMES:
Complete Response (CR) | Up to 5 years
  CR will be determined for each subject as a binary variable indicating whether the achieved a best overall response to induction therapy of CR or better
Best Response | Up to 5 years
  The best overall response will be determined as an ordered categorial variable indicating the subject's best response at any point along the treatment continuum.
Very Good Partial Response (VGPR) | up to 5 year
  will be determined for each subject as a binary variable indicating whether the achieved a best overall response to induction therapy of VGPR or better.
Overall Response | up to 5 years post treatment discontinuation
  The best overall response will be determined as an ordered categorial variable indicating the subject's best response at any point along the treatment continuum
MRD Negative | Up to 5 years
  . Minimal residual disease (MRD) (via NGF 10-5 and 10-6) will be determined for each subject after suspected CR for Phase I subjects and at the following timepoints for Phase II subjects: after induction therapy, after ASCT, and after 12 cycles of maintenance therapy (post Cycle 18visit) and every 12 months post Cycle 18 sample.
Time to First Response (TTFR) | up to 30 days post treatment discontinuation
  TTFR will be calculated for all subjects achieving an sCR, CR, VGPR, or PR. This will be defined as the time from initiation of belantamab mafodotin-containing protocol directed induction therapy to the time of first disease assessment indicating either sCR, CR, VGPR or PR
Time to Best Response (TTBR) | up to 30 days post treatment discontinuation
  Time to best response will be calculated for all subjects achieving an sCR, CR, VGPR or PR. This will be defined as the time from initiation of belantamab mafodotin-containing protocol directed induction therapy to the time of best disease assessment indicating either sCR, CR, VGPR or PR.
Time to Progression (TTP) | Up to 5 years
  TTP is defined as the duration of time from enrollment to the study (treatment start date) to first occurrence of progressive disease
Duration of Response (DoR) | Up to 5 years post treatment response
  DoR will be calculated for each subject achieving a PR or better and will be calculated from the time of the first assessment that identified response until disease progression or death.
Overall Survival (OS) | Up to 8 years
  OS is defined as the duration from enrollment to the study (treatment start date) to the date of death from any cause.
Progression Free Survival (PFS) | Up to 8 years
  PFS is defined as the duration of time from enrollment to the study (treatment start date) to first occurrence of either progressive disease or death (from any cause), whichever comes first.

OTHER OUTCOMES:
Safety - Serious Adverse Events (SAEs) | Up to 4-8 weeks post treatment discontinuation
  The SAE variable will be determined for each subject as a binary variability indicating whether or not subject experienced a protocol-defined SAE.
Safety - Adverse Events (AEs) | Up to 4-8 weeks post treatment discontinuation
  The AE variable will be determined for each subject as a binary variability indicating whether or not subject experienced an AE per CTCAE V5.0.
Safety - Adverse Events of Special Interest (AESIs) | Up to 4-8 weeks post treatment discontinuation
  The AESI variable will be determined for each subject as a binary variability indicating whether or not subject experienced a protocol-defined AESI.
Translational Research - PFS and OS | Up to 8 years
  Describe subject outcomes of progression free survival and overall survival for MRD concordant and discordant cases
Translational Research - MRD Status | Up to 8 years
  Compare MRD status concordance between NGF and QiP mass spectrometry
Translational Research - BCMA expression | Up to 8 years
  Assess BCMA (B Cell Maturation Antigen) expression by plasma cells prior to therapy and at relapse using formalin-fixed paraffin embedded (FFPE) bone marrow biopsies.
Translational Research - Immunologic Profiles | Up to 8 years
  Establish peripheral blood and bone marrow immunologic profiles throughout therapy.
Translational Research - plasma BCMA expression | Up to 8 years
  Correlate plasma cell BCMA (B Cell Maturation Antigen) expression with Progression Free Survival (PFS) and Overall Survival (OS).
Translational Research - serum BCMA concentration | Up to 8 years
  Correlate serum cell sBCMA (serum B Cell Maturation Antigen) concentration with Progression Free Survival (PFS) and Overall Survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Shebli Atrash, MD, MS, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No